CLINICAL TRIAL: NCT06083662
Title: Phase II Basket Trial to Evaluate Safety and Efficacy of Neratinib, an Irreversible Tyrosine Kinases Inhibitor of EGFR, ERBB2 and ERBB4 Receptors and Trastuzumab Biosimilar (Herzuma®) in Patients with HER2 Mutated Advanced Solid Cancers
Brief Title: Neratinib and Trastuzumab Biosimilar in Patients with HER2 Mutated Advanced Solid Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, Park, In Hae, MD, PhD, Korea University Guro Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL20-17
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Cancer; HER2 Gene Mutation
MeSH Terms: conditions — Neoplasm Metastasis | interventions — neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A arm (Experimental): Neratinib + herzuma
  Interventions: Drug: Neratinib Maleate

INTERVENTIONS:
Drug: Neratinib Maleate — * neratinib 240mg po daily
  * herzuma 8mg/kg (loading) --> 6mg/kg q3w
  Other Names: Herzuma

SUMMARY:
Prospective, Basket, Open-label, Multi-dose, Single-arm, Simon's two-stage, Multi-center trial

Study drug : neratinib + herzuma (trastuzumab biosimilar)

DETAILED DESCRIPTION:
1. Primary objective Evaluate overall response rate (ORR) in HER2 mutated advanced solid cancer patients based on RECIST v1.1
2. Secondary objectives

(1) Evaluate clinical benefit rate (CBR) (2) Evaluate duration of response (DOR) (3) Evaluate progression free survival (PFS) (4) Evaluate overall survival (OS) (5) Evaluate compliance with oral administration 3) Safety evaluation

1. Evaluate the overall safety of the test drug
2. Evaluate the predefined adverse event (diarrhea)

ELIGIBILITY:
Inclusion Criteria:

* Patients who voluntarily decide to participate and give written consent after hearing the explanation of the clinical trial and investigational drugs.
* Adult men and women over 19 years old.
* Histological or cytological confirmed advanced solid tumor and confirmed to have HER2 known oncogenic mutations in tumor DNA by K-master panel test using tumor tissues or circulating tumor DNA in blood.
* Patients having at least 1 or more than 1 measurable lesion according to RECIST v 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status 0~2.
* Patients whose life expectancy is more than 6 months.
* Metastatic/progressive solid cancer patients who have received one or more than one standard treatment or do not have any treatment option.
* Patients who have agreed to provide plasma/blood samples, the most recent metastatic/progressive tumor sample or new tumor biopsy for gene sequencing and other biomarker analysis.

Exclusion Criteria:

* Patients who received radiotherapy or surgical treatment within 2 weeks prior to the initiation of investigational product.
* Patients having symptomatic brain metastasis who needs treatment. Patients with stable brain metastasis who need no treatment including steroid are eligible
* Inappropriate HER2 mutation (e.g., non-Hot Spot mutation, variant of unknown siginificance, subclonal mutation, premature STOP codon or the Frame Shift mutation).
* Patients having difficulties in swallowing tablets.
* Patients with toxicities of prior treatment which are not recovered to baseline level or ≤ Grade 1.
* Inadequate organ functions:

  1. Hemoglobin (Hemoglobin) < 8 .0g / dL
  2. Absolute neutrophil count (ANC) < 1. 0 x10 ³ per mm³
  3. Platelet count < 100 x10⁹/L (100 ,000/ mm³)
  4. Total bilirubin > 1.5 x upper normal limits (UNL), (exclude Gilbert's syndrome)
  5. Alanine aminotransferase (ALT) or aspartate amino transferase (AST) > 3 x upper normal limits (UNL) (in case of liver and bone metastases > 5 x ULN)
  6. Serum creatinine >1.5 x upper normal limits (UNL) or < eGFR 30 mL/min/1.73 m² 7) Left ventricle ejection fraction <50% by multi-gate obtaining method scan (MUGA) or echocardiogram.

  8) Chronic gastrointestinal disorders of which a main symptom is diarrhea (e.g., Crohn's disease, malabsorption, or grade 2 or more than grade 2 diarrhea according to the NCI CTCAE version 5.0 regardless of etiology).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
overall response rate (ORR) | at 6 months
  ORR according to RECIST v1.1

SECONDARY OUTCOMES:
clinical benefit rate, CBR | at 6 months
  CR+PR + SD more than 12 weeks
median duration of response, DOR | at 6 months
  DOR is related to the quality of life and is one of the methods for evaluating tumor response approved by pharmaceutical regulatory agencies
median progression free survival, PFS | at 6 months
  from enrollment to disease progression, death or withdrawal
safety profiles | at 6 months
  safety profiles according to CTCAE 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Korea university Guro hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No